CLINICAL TRIAL: NCT05785403
Title: Co-designing Improvements in Care and Self-care Opportunities for Scleroderma Digital Ulcers With Patients and Clinicians
Brief Title: Co-designing Digital Ulcers Opportunities With Patients and Clinicians
Acronym: CoDUo
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: King's College London (Other)
Collaborators: Royal Free Hospital NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: IRAS 320344
Record Dates: First submitted 2023-03-06; First posted 2023-03-27 (Actual); Last update posted 2023-03-27 (Actual); Status verified 2023-03

CONDITIONS: Scleroderma; Scleroderma Associated Digital Ulcer; Digital Ulcer
MeSH Terms: conditions — Scleroderma, Diffuse; digital ulcers

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
Scleroderma (SSc) is a rare crippling chronic disease associated with damage of the blood vessels and hardening of connective tissue. It has quite a number of complications including ulcers to the fingers and toes (digital ulcers).

Digital ulcers (DU) are a frequent challenge in patients with SSc (PwSSc), as they approximately affect more than half of these patients. Care received by PwSSc DU is varied. Patients with three or more ulcers are considered to have severe disease therefore these patients usually receive expensive treatments and referred to specialist SSc clinics, while those with less ulcers may not receive the same treatments, and only see their general practitioner or local rheumatologist or left to their own means. Resulting in patients developing their own DU managing practices which may be good and some not.

Currently, no research has fully identified the needs of PwSSc DU and self-care interventions to support them are lacking. The extent to which DU support needs are met by non-specialist health professionals is unknown. There is lack of literature in co-designing interventions with patients in SSc DU. Developing interventions and pathways for managing DU with patients and healthcare professionals (HCP) will enhance DU care and lessen the burden for the affected patients, a qualitative study is required.

Aim The aim of this research is to co-design self-care opportunities and develop improvements in DU care.

Objectives

1. to explore how patients with SSc DU are currently managed
2. to understand how they currently manage their ulcers and their healthcare needs.
3. to collaboratively co-design self-care opportunities and improvements in care.

Study Methods Experience-based co-design (EBCD) qualitative methodology will be used to conduct the study. 10 HCP and 12-15 PwSSc DU will be invited to participate in consultation observations. Followed by individuals interviews for the HCP and PwSSc DU care and perceptions on unmet needs. The results will inform collaborative co-designing and development of interventions with patients and HCP. The same participants will also be invited to participate in three workshops involving designing, discussion, refinement and finalisation of the interventions. The interventions developed will be ready to be tested or being evaluated once they have been put in place..

ELIGIBILITY:
Inclusion Criteria:

* Healthcare Professionals who see People with SSc DU
* Patients ≥18 years old
* Patients fulfilling the 2013 American College of Rheumatology -European Alliance of Associations for Rheumatology classification criteria for SSc
* Patients with a history of previous DU or current DU regardless the number of ulcers
* Participants able to provide informed written consent

Exclusion Criteria:

* Healthcare professionals who see patients with rheumatological conditions but not SSc
* Patients aged below ≤18 years old
* Patients with DU, however without diagnosis of SSc
* Patients diagnosis of SSc who have never had DU
* Participants who do not speak English, hence cannot provide informed consent, or participant in interviews

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Healthcare professionals who see patients with SSc DU Patients diagnosed with SSc DU
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2023-06 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Qualitative co-designed self-care interventions and improved DU care services | 12 months
  Patients and healthcare professionals will be recruited for consultation observations and interview to find out DU care needs. The qualitative analysis will lead to jointly co-designing self-care interventions and DU care service re-design.